CLINICAL TRIAL: NCT00795847
Title: The Efficacy and Safety of Losartan/Hydrochlorothiazide Combination Drug (Preminent) in Patients With Morning Hypertension
Brief Title: Morning Hypertension and Preminent Therapy Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kurume University (Other)
Responsible Party: Tsutomu Imaizumi/Chair of Cardio-vascular Medicine Kurume University, Cardio-vascular Medicine Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KurumeU-08058
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
Keywords: Hypertensive patients with morning hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Preminent (Experimental): Patients with blood pressure self-measurement-proven morning hypertension are treated with Preminent 1T qd for 3 months.
  Interventions: Drug: Preminent (losartan/hydrochlorothiazide combination drug)
- 2. High-dose losartan (Active Comparator): Patients with blood pressure self-measurement-proven morning hypertension are treated with losartan 100 mg qd for 3 months.
  Interventions: Drug: Preminent (losartan/hydrochlorothiazide combination drug)

INTERVENTIONS:
Drug: Preminent (losartan/hydrochlorothiazide combination drug) — Preminent 1T qd (Arm 1) or losartan 100 mg (Arm 2) was given for 3 months.

SUMMARY:
It is difficult to control morning hypertension in practical clinical situation. Angiotensin receptor blocker (ARB) and thiazide are suggested to be effective to maintain the antihypertensive effects for 24 hours. However, monotherapy sometimes is not enough to control blood pressure level in the next morning and there are little evidence of the combination therapy for morning hypertension. The investigators hypothesized that a losartan 50 mg/hydrochlorothiazide 12.5 mg combination drug, Preminent, is effective and safe for controling morning hypertension, compared with high-dose of losartan 100 mg, in Japanese. Patients with morning hypertension were randomized to preminent treatment group or high-dose losartan treatment group. The efficacy and safety were compared after 3-month treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of outpatients with morning hypertension (135/85 mmHg)
* Under treatment with any antihypertensive agents

Exclusion Criteria:

* Poorly controlled hypertension (DBP>120 mmHg)
* Poorly controlled diabetes (HbA1c>9.0%
* Gout or hyperuricemia (UA>8.0 mg/dL)
* Serum Cr>2.0 mg/dL
* Serum K>5.5 mmol/L
* Liver dysfunction (ALT>90 IU/L and/or g-GTP>14o IU/L)
* Secondary hypertension
* Patients who have contraindication for losartan and/or thiazide diuretics

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure level in the morning by blood pressure self-measurement | 3 months

SECONDARY OUTCOMES:
Serum levels of potassium, BUN, Creatinine, Uric acid, and Brain natriuretic peptide | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Imaizumi, MD, PhD, Study Chair — Kurume University; Hisashi Kai, MD, PhD, Principal Investigator — Kurume University
Locations (1):
- Cardio-vascular Medicine, Kurume University, Kurume, Fukuoka, Japan